CLINICAL TRIAL: NCT01197612
Title: Nasal Packing as a Drug Delivery System Postoperatively in Chronic Sinusitis With Polyposis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: American Rhinologic Society (Other)
Responsible Party: Principal Investigator, Garrett Griffin, Resident/Research Fellow, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: HUM00029273
Record Dates: First submitted 2010-08-30; First posted 2010-09-09 (Estimated); Results first posted 2018-05-29 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-04

CONDITIONS: Chronic Sinusitis; Polyposis
MeSH Terms: interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm; nostrils as experimental and comparator (Other): each subject serves as their own control with one nostril being treated with pulmicort and one not
  Interventions: Drug: pulmicort

INTERVENTIONS:
Drug: pulmicort — applied to nasal packing after surgery
  Other Names: budesonide

SUMMARY:
That high-dose steroid applied to the nasal cavity immediately post-operatively will improve olfaction and healing following endoscopic sinus surgery.

ELIGIBILITY:
Inclusion Criteria:

* hyposmia and nasal obstruction for >12 weeks
* bilateral nasal polyposis
* candidate for surgery

Exclusion Criteria:

* immunocompromised
* non-English speaking
* prisoner
* pregnant/lactating
* will not attend follow up appointments

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Garrett R Griffin, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 23 participants who consented, data is only available for 20. Two never had surgery, and so were not "assigned" at all.
Period: Overall Study
Arm/Group | Single Arm; Nostrils as Experimental and Comparator
Started | 18
Week 3 | 16
Returned for Week 24 | 6
Completed | 6
Not Completed | 12

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm; Nostrils as Experimental and Comparator
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Olfaction
Description: will be measured with the University of Pennsylvania Smell Identification Test (UPSIT), whose scores range from 0 to 40, where 0 is the inability to smell anything and 40 is perfect smell identification
Time Frame: 3 weeks post-operation
Population: Of sixteen participants at the three week mark, one participant's data was unable to be unblinded accurately, and one participant had no UPSIT scores taken, leaving an analysis population of 14,
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Treated Nostril (Pulmicort); Untreated Nostril (no Pulmicort): each subject serves as their own control with one nostril being treated with pulmicort and one not
  pulmicort: applied to nasal packing after surgery
Arm/Group | Treated Nostril (Pulmicort) | Untreated Nostril (no Pulmicort)
Number analyzed (Participants) | 14 | 14
units on a scale | 20.2 [8 to 36] | 19.8 [6 to 37]

2. Secondary Outcome: Sinonasal Health
Description: will be assessed with the Perioperative Sinus Endoscopy score (POSE), a 20 point scale where 0 is no sinus challenges and 20 represents the greatest blockage.
Time Frame: 3 weeks post operation
Population: unblinding could not be done on one person accurately, so only 15 rather than 16 people's data could be analyzed
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Placebo Treated Nostril (no Pulmicort): each subject serves as their own control with one nostril being treated with pulmicort and one not
  pulmicort: applied to nasal packing after surgery
Arm/Group | Treated Nostril (Pulmicort) | Placebo Treated Nostril (no Pulmicort)
Number analyzed (Participants) | 15 | 15
units on a scale | 4.5 [1 to 10] | 4.7 [0 to 10]

3. Secondary Outcome: Olfaction
Description: Scored with the University of Pennsylvania Smell Identification Test, whose scores range from 0 to 40, where 0 is the inability to smell anything and 40 is perfect smell identification
Time Frame: 24 weeks post operation
Population: Of six participants remaining at 24 weeks, one participant's data could not be accurately unblinded leaving analysis of 5
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Placebo/Untreated Nostril (no Pulmicort): each subject serves as their own control with one nostril being treated with pulmicort and one not
  pulmicort: applied to nasal packing after surgery
Arm/Group | Treated Nostril (Pulmicort) | Placebo/Untreated Nostril (no Pulmicort)
Number analyzed (Participants) | 5 | 5
units on a scale | 20.4 [9 to 37] | 20 [7 to 38]

4. Secondary Outcome: Sinonasal Health
Description: Assessed with Perioperative Sinus Endoscopy (POSE) score
Time Frame: 24 weeks post operation
Population: Of six participants at 24 weeks, one's data was unable to be unblinded accurately, leaving an analysis population of 5 participants
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Treated Nostril (Pulmicort) | Untreated Nostril (no Pulmicort)
Number analyzed (Participants) | 5 | 5
units on a scale | 5.6 [0 to 11] | 5.6 [2 to 11]

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Single Arm; Nostrils as Experimental and Comparator
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

LIMITATIONS AND CAVEATS:
This was a pilot study with less enrollment than desired and poor rate of completion with only 5 participants completing the full 24 week trial. This study could be done on a larger/similar scale with some additional useful data obtained.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No